CLINICAL TRIAL: NCT03320720
Title: Evaluation of Home Treatment for Acute Psychiatric Care of the Psychiatric University Hospital Zurich (Switzerland)
Brief Title: Evaluation of Home Treatment for Acute Psychiatric Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Matthias Jäger, PD Dr. med., Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HT201701349
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Treatment (Experimental): Patients with acute mental illness are treated at their houses by a mobile and multiprofessional care team instead of being treated as inpatients if their medical condition permits.
  Interventions: Other: Home Treatment
- Treatment-as-usual (Active Comparator): Patients with acute mental illness are treated as inpatients in a psychiatric clinic.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Other: Home Treatment — Patients with acute mental illness in need of inpatient care are treated at their houses by a mobile and multiprofessional care team if their health condition permits.
  Arms: Home Treatment
Other: Treatment-as-usual — Patients with acute mental illness in need of inpatient care are treated in a psychiatric clinic.
  Arms: Treatment-as-usual

SUMMARY:
The study's goal is to evaluate whether home treatment is an effective and efficient alternative to inpatient care for people with acute mental illness. Patients who meet the study's inclusion criteria are randomly assigned to either the condition home treatment or inpatient care (treatment-as-usual), during one year. Following two years, the two treatment modalities will be analyzed in terms of inpatient days, cost effectiveness, rehospitalization rate, severity of symptoms and sociodemographics.

DETAILED DESCRIPTION:
The study's goal is to evaluate whether home treatment is an effective and efficient alternative to inpatient care for people with acute mental illness. Therefore, psychiatric patients in need of hospitalization who meet the study's inclusion criteria are randomly assigned to either the condition home treatment or inpatient care (treatment-as-usual) during one year. Home treatment patients are visited by a mobile and multiprofessional care team at their homes. Additionally, patients without a health insurance for home treatment and patients who are directly assigned to home treatment are included in separate study groups. Following two years, it will be checked whether home treatment leads to a reduction of inpatient days as a primary outcome. Further outcomes such as cost effectiveness, rehospitalization rate, severity of symptoms and sociodemographics will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Need for acute psychiatric inpatient care
* Residence in Zurich city
* Health insurance for Home Treatment

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Inpatient days | 2 years follow-up
  Number of inpatient days per patient

SECONDARY OUTCOMES:
Total days in treatment | 2 years follow-up
  Total days in Treatment per patient = inpatient and home treatment
Treatment costs | 2 years follow-up
  Calculated direct treatment costs
Rehospitalization rate | 2 years follow-up
  Number of rehospitalizations per patient and duration until rehospitalization
Adverse events | 2 years follow-up
  e.g. suicide or attempted suicide
Global Assessment of Functioning Scale (GAF) | 2 years follow-up
  Scale measures social, occupational and psychological functioning and ranges from 0 to 100 (higher values mean better outcome).
Health of the Nation Outcome Scale (HoNOS) | 2 years follow-up
  Scale measures the severity of symptoms and ranges from 0 to 48 (higher values mean worse outcome).
Clinical Global Impression Scale (CGI) | 2 years follow-up
  Scale measures the severity of symptoms, global improvement and therapeutic response and ranges from 0 to 7 (higher values mean worse outcome).
Patients' satisfaction | 2 years follow-up
  Patients' satisfaction assessed by the official questionnaire of the national association of the quality development in hospitals (ANQ)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Jäger, MD, Principal Investigator — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No